CLINICAL TRIAL: NCT04438083
Title: A Phase 1 Dose Escalation and Cohort Expansion Study of the Safety and Efficacy of Allogeneic CRISPR-Cas9-Engineered T Cells (CTX130) in Subjects With Advanced, Relapsed or Refractory Renal Cell Carcinoma With Clear Cell Differentiation
Brief Title: A Safety and Efficacy Study Evaluating CTX130 in Subjects With Relapsed or Refractory Renal Cell Carcinoma (COBALT-RCC)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Patients to be followed up in the CRSP-ONC-LTF study
Sponsor: CRISPR Therapeutics AG (Industry)
Responsible Party: Sponsor
Organization: CRISPR Therapeutics (Industry)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CRSP-ONC-003
Record Dates: First submitted 2020-06-16; First posted 2020-06-18 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Renal Cell Carcinoma
Keywords: CAR T; Allogeneic; Renal cell carcinoma; Renal cell carcinoma with clear cell differentiation; CRISPR-Cas9
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CTX130 (Experimental): Administered by IV infusion following lymphodepleting chemotherapy.
  Interventions: Biological: CTX130

INTERVENTIONS:
Biological: CTX130 — CTX130 CD70-directed T-cell immunotherapy comprised of allogeneic T cells genetically modified ex vivo using CRISPR-Cas9 gene editing components.

SUMMARY:
This is a single-arm, open-label, multicenter, Phase 1 study evaluating the safety and efficacy of CTX130 in subjects with relapsed or refractory renal cell carcinoma.

DETAILED DESCRIPTION:
The study may enroll approximately 107subjects in total.

ELIGIBILITY:
Abbreviated Inclusion Criteria:

1. Age ≥18 years and body weight ≥42 kg.
2. Unresectable or metastatic RCC that has exploited standard of care treatment.
3. Karnofsky performance status (KPS) ≥80%.
4. Adequate renal, liver, cardiac, and pulmonary organ function.
5. Female subjects of childbearing potential and male subjects must agree to use acceptable method(s) of contraception from enrollment through at least 12 months after CTX130 infusion.

Abbreviated Exclusion Criteria:

1. Prior treatment with any anti-CD70 targeting agents.
2. Prior treatment with any CAR T cells or any other modified T or natural killer (NK) cells.
3. History of certain central nervous system (CNS), cardiac or pulmonary conditions.
4. Active HIV, hepatitis B virus or hepatitis C virus infection.
5. Previous or concurrent malignancy, except treated with curative approach not requiring systemic therapy and in remission for >12 months, or any other localized malignancy with low risk of developing into metastatic disease.
6. Primary immunodeficiency disorder or active autoimmune disease requiring steroids and/or other immunosuppressive therapy.
7. Prior solid organ transplantation or bone marrow transplant.
8. Pregnant or breastfeeding females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2020-06-16 (Actual); Primary Completion 2024-10-08 (Actual); Study Completion 2024-10-08 (Actual)

PRIMARY OUTCOMES:
Part A (dose escalation): Incidence of adverse events | From CTX130 infusion up to 28 days post-infusion
  Adverse events defined as dose-limiting toxicities
Part B (cohort expansion): Objective response rate | From CTX130 infusion up to 60 months post-infusion]
  Objective response rate per Response Evaluation Criteria In Solid Tumors (RECIST) v1.1

SECONDARY OUTCOMES:
Progression Free Survival | From date of CTX130 infusion until date of disease progression or death due to any cause, assessed up to 60 months
Overall Survival | From date of CTX130 until date of death due to any cause, assessed up to 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Alissa Keegan, MD, Study Director — CRISPR Therapeutics
Locations (7):
- United States (4):
  - Research Site 2, Duarte, California
  - Research Site 5, Hartford, Connecticut
  - Research Site 4, Houston, Texas
  - Research Site 3, Salt Lake City, Utah
- Research Site 1, Melbourne, Victoria, Australia
- Research Site 6, Toronto, Ontario, Canada
- Research Site 7, Amsterdam, North Holland, Netherlands

REFERENCES:
- [Derived] Dewulf J, Flieswasser T, Delahaye T, Vangestel C, Miranda A, de Haard H, Jacobs J, Smits E, Van den Wyngaert T, Elvas F. Site-specific 68Ga-labeled nanobody for PET imaging of CD70 expression in preclinical tumor models. EJNMMI Radiopharm Chem. 2023 Apr 24;8(1):8. doi: 10.1186/s41181-023-00194-3. PMID 37093350